CLINICAL TRIAL: NCT04953143
Title: LiverPAL: A Pilot Study of Inpatient Palliative Care for Patients With Advanced Liver Disease
Acronym: LiverPal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Association for the Study of Liver Diseases (Other)
Responsible Party: Principal Investigator, Nneka nnaoke Ufere, Instructor in Internal Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021P001402
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot (Experimental): Inpatient longitudinal palliative care intervention that includes the following domains:
  * Therapeutic relationship: Developing trust and credibility with patients and their families
  * Symptom management: Proactive symptom management for common advanced liver disease symptoms including pain, fatigue, anorexia, breathlessness, depression and anxiety
  * Coping with illness: Introduction of strategies to improve adjustment and meaning in life; bolstering caregiver coping
  * Prognostic awareness and illness understanding: Assessing patients' level of prognostic awareness and discussing strategies to help patients cope with uncertainty
  * Treatment decision-making: Supporting patients and caregivers in their medical decision-making and assessing their values in decision-making
  * End-of-life care: Review/discuss selection of healthcare proxy, preferences for end-of-life care
  Interventions: Behavioral: LiverPal Intervention

INTERVENTIONS:
Behavioral: LiverPal Intervention — Inpatient longitudinal palliative care intervention
  - Patients will complete baseline assessments and will be followed by the palliative care clinicians delivering the LiverPal intervention during each of their hospitalizations over a 3 month period
  LiverPal intervention domains include the following:
  * Therapeutic relationship
  * Symptom management
  * Coping with illness
  * Prognostic awareness and illness understanding
  * Treatment decision-making
  * End-of-life care

SUMMARY:
Frequently patients with advanced liver disease experience physical and emotional symptoms during their hospitalization that can may cause a level of discomfort to both the patient and the family members that surround them.

This study involves the early introduction of a team of clinicians that specialize in the lessening (palliation) of many of these discomforting symptoms. This team of clinicians is called the palliative care team and they focus on ways to improve pain and other symptom management and to assist patients and their families in coping with the physical, emotional and social issues associated with a diagnosis of advanced liver disease. The team consists of physicians and advance practice nurses who have been specially trained in the care of patients facing serious illness and their caregivers.

The investigators are studying the feasibility of delivering this program, the acceptability and satisfaction with the program, and changes in the quality of life, illness understanding, and symptoms of hospitalized patients who receive the program and their caregivers. The study will use a series of questionnaires to measure the study participants' quality of life, physical symptoms, illness and prognostic understanding, and mood. Study questionnaires will be completed in the hospital, home or clinic. Qualitative interviews will be conducted with hepatology and palliative care clinicians as well as patients and caregivers.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Adult (≥ 18 years old) with advanced liver disease defined as cirrhosis complicated by one of the following (new or ongoing) clinically-evidence decompensating events

   1. Ascites (requiring diuretics or large volume paracenteses)
   2. Hepatic encephalopathy (requiring medical therapy)
   3. History of variceal bleed episode within 1 year of enrollment
2. Admitted to the general medicine service
3. Ability fo communicate in English and provide informed consent
4. Have a score ≥ 7 on the Short Portable Mental Status Questionnaire

Patient Exclusion Criteria:

1. Patients with severe hepatic encephalopathy or any other comorbid condition which the primary medical team believes prohibits compliance with study procedures
2. Patients with advanced malignancies being treated with palliative intent
3. Patients already receiving specialty palliative care and/or hospice care

Caregiver Eligibility Criteria

1. A relative or friend of eligible patient, who lives with them and has in-person contact with them at least twice per week
2. Verbally fluent in English or able to complete questionnaires with the help of an interpreter
3. Age 18 or older

Clinician Selection: All palliative care clinicians who deliver the LiverPal intervention will participate in qualitative interviews. Inpatient clinicians who provided direct care to enrolled patients in either the inpatient or outpatient setting will also be eligible to participate in the qualitative interviews.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
LiverPal intervention refinement | Time Frame: Up to 1 year
  The investigators will conduct qualitative interviews with the patients and caregivers enrolled in the open pilot phase as well as LiverPal clinicians to elicit stakeholder feedback on the intervention. The qualitative component of the exit interviews will explore 1) patients', caregivers' and clinicians' perceptions of the acceptability and content of LiverPal; 2) any barriers or challenges to providing or receiving LiverPal; and 3) suggested modifications to LiverPal to improve its delivery in the inpatient setting

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No